CLINICAL TRIAL: NCT02122874
Title: Percutaneous Electric Neurostimulation of Dermatome T7 Improves Glycemic Profile in Obese and Typo 2 Diabetic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, MD, PhD, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-003
Record Dates: First submitted 2014-04-18; First posted 2014-04-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes Mellitus Type 2 in Obese; Type 2 Diabetes Mellitus With Features of Insulin Resistance
Keywords: Percutaneous neurostimulation; dermatome T7, type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Diet (Active Comparator): The patients follow only a 1200 Kcal diet
  Interventions: Device: Percutaneous Neurostimulation (PENS) of dermatome T7; Other: 1200 Kcal diet
- Diet +PENS dermatome T7 (Experimental): The patients undergo PENS of dermatome T7 and follow a 1200 Kcal diet
  Interventions: Device: Percutaneous Neurostimulation (PENS) of dermatome T7

INTERVENTIONS:
Device: Percutaneous Neurostimulation (PENS) of dermatome T7 — The patients undergo PENS of dermatome T7 and follow a 1200 Kcal diet
Other: 1200 Kcal diet
  Arms: Diet

SUMMARY:
Percutaneous neurostimulation of dermatome T7 increases Insulin segregation by the apancreas and improves glycemic profile in diabetic patients

ELIGIBILITY:
Inclusion Criteria:

* BMI>30 Kg/m2
* Type 2 diabetes mellitus
* Treatment with Metformin

Exclusion Criteria:

* Under insulin treatment
* Endocrinological disorders causing diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Serum glucose levels (mg/dl) | Baseline and 12 weeks after beginning the therapy
  Serum glucose levels will be recorded will be recorded at baseline and 12 weeks after beginning the treatment. Measurement units will be mg/dl.

SECONDARY OUTCOMES:
Homeostasis model assessment (HOMA) | Baseline and 12 weeks after beginning the therapy
  Insulin resistance will be recorded by the Homeostasis model assessment (HOMA). The calculation formula is: Serum Glucose x Serum Insulin / 405

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital Elche, Elche, Alicante, Spain